CLINICAL TRIAL: NCT05716802
Title: Dance/Movement Therapy for Improving Bone Mineral Density in Long-term Patients With Schizophrenia: a Randomized Controlled Trial
Brief Title: Dance/Movement Therapy for Bone Mineral Density in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hebei Province Veterans Hospital (Other Government)
Responsible Party: Principal Investigator, Hengyong Guan, Principal Investigator, Hebei Province Veterans Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: xmh123
Record Dates: First submitted 2023-01-29; First posted 2023-02-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dance/movement therapy (DMT), twice a week, 12 weeks, (Active Comparator): The multiple-session DMT intervention was applied to participants twice a week as a total of 24 sessions of 60 minutes over three months. The DMT intervention protocol was developed based on the therapist's experience, the theoretical frameworks, and the DMT approach described in a previous study (Bryl and Goodill 2019).
  Interventions: Behavioral: dance/movement therapy
- Treatment as usual (TAU), twice a week, 12 weeks, (Placebo Comparator): The TAU group sessions were conducted by the licensed professional employed at the hospital. The patients received regular daily antipsychotic medication and supportive psychotherapy once a week. They also participated in daily activities from Monday to Friday for at least two hours each day, including indoor activities (watching TV, playing games, playing poker) and outside activities (walking and doing radio gymnastics).
  Interventions: Behavioral: treatment as usual

INTERVENTIONS:
Behavioral: dance/movement therapy — dance/movement therapy plus treat as usual
  Arms: dance/movement therapy (DMT), twice a week, 12 weeks,
Behavioral: treatment as usual — The patients received regular daily antipsychotic medication and supportive psychotherapy once a week. They also participated in daily activities from Monday to Friday for at least two hours each day, including indoor activities (watching TV, playing games, playing poker) and outside activities (walking and doing radio gymnastics).
  Arms: Treatment as usual (TAU), twice a week, 12 weeks,

SUMMARY:
Fractures are common accidents for long-term hospitalized patients with schizophrenia (SZ) in psychiatric hospitals, and once they occur, patients usually endure the pain of fractures for a long time. Accumulating evidence has supported implementing dance/movement therapy (DMT) as a promising intervention for patients with SZ. However, no study has been conducted to investigate its role in balance ability and metabolic parameters in SZ. This study was designed to investigate the treatment outcome of a 12-week DMT intervention on bone mineral density, balance ability, and metabolic profile in patients with SZ using a randomized, controlled trial design.

DETAILED DESCRIPTION:
Schizophrenia (SZ) is a chronic, severe psychiatric disorder that affects approximately 1% of the population. The psychiatric symptoms and high rate of relapse of SZ can significantly impair cognitive and social functioning, including problem-solving skills, interpersonal relationships, and work performance. Moreover, individuals with SZ usually have higher disability and premature mortality rates compared to the general population. Falls are a common concern in hospital settings, with studies reporting a fall rate between three and five falls per 1000 bed days. Osteoporosis and its precursors, e.g. osteopenia and low bone mineral density (BMD), have been reported in chronic patients with SZ and were strong predictors for subsequent falls and fractures in psychiatric hospitals.

Dance/movement therapy (DMT), as one of the creative arts therapies, is an emerging therapy for the rehabilitation of patients with SZ in recent years. DMT therapy uses dance activities and body movements to enhance well-being, mood, and quality of life. DMT therapy uses movement, dance, and interpersonal communication to explore a person's emotional, cognitive, social, and physical integration, enabling patients to enhance self-expression, accept and reconnect with their bodies, and strengthen their fitness. The patients share their emotions, concerns, and coping strategies with others through dance/movement. It can be applied to individuals of all ages, races, and genders and can be efficacious in individuals who experience losses in social, physical, and psychological functions. DMT has also been used to improve the cognition and social function of patients with mental diseases in psychiatric hospitals. In particular, a few studies have reported a critical role of DMT intervention in negative symptoms in chronic patients with SZ. However, there is still a lack of evidence that whether DMT is an effective therapy to increase the mean bone mineral density and reduce the risk of fractures due to falls in long-term hospitalized patients with SZ.

In the present study, the investigators hypothesized that DMT intervention was effective to increase BMD and balance ability and decrease the metabolic parameters in long-term hospitalized male veterans with SZ as compared to the control group. They also examined whether DMT intervention can significantly change BMI, the levels of lipid profile, and serum calcium in patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of schizophrenia using the DSM-V;
* male veterans, aged 40 to 60 years with a disease duration of 5 years or more and a long-term hospitalization of 3 years or more;
* ability to understand Mandarin Chinese;
* legally eligible to sign an informed consent form;
* current antipsychotic medication stability for more than 2 years;
* reduced bone mass, osteoporosis, and severe osteopenia after bone density analysis;
* no comorbid serious physical illness and physical impairments and can cooperate with nurses to complete the general intensity of activity training;
* consent for pre- and post-session interviews.

Exclusion Criteria:

1) substance dependence or abuse; 2) hypercalcemia and hyperuricemia; 3) history of kidney stones or renal calculi; 4) lower limb injury and motor dysfunction, and inability to complete DMT intervention for various reasons.

-

Ages: 40 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-07-07 (Actual); Primary Completion 2022-01-12 (Actual); Study Completion 2022-07-12 (Actual)

PRIMARY OUTCOMES:
Bone mineral density measurement | week 12
  The primary outcome measure was the BMD of patients recruited, which was assayed by an Erik AKDX-09W-1 bone density device (Shenzhen Ekere Electric Co.). The test was performed using the dual-energy X-ray absorptiometry method. Measurements were done at the distal end of the flexor bone of the patient's left forearm for fan beam and line scan, which were reviewed by an experienced radiologist who was blinded to the clinical and pharmacological characteristics and randomization of the patients.

SECONDARY OUTCOMES:
panss scale | week 12
  THE POSITIVE AND NEGATIVE SYNDROME SCALES. The minimum and maximum values are 28 and 198. Higher scores mean a worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Hengyong Guan, Dr., Study Director — Hebei Province Veterans Hospital
Locations (1):
- DMT, Baoding, Hebei, China

IPD SHARING:
Plan to Share IPD: No